CLINICAL TRIAL: NCT03893071
Title: An Open-Label Extension Study of the Long-Term Safety and Efficacy of Intravenous Trappsol® Cyclo (HP-β-CD) in Patients With Niemann-Pick Disease Type C (NPC-1)
Brief Title: Open-Label Study of Long-Term Safety and Efficacy of Intravenous Trappsol Cyclo (HPβCD) in Niemann-Pick Disease Type C
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cyclo Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTD-TCNPC-102
Record Dates: First submitted 2019-02-20; First posted 2019-03-28 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-02

CONDITIONS: Niemann-Pick Disease, Type C1
MeSH Terms: conditions — Niemann-Pick Disease, Type C

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Hydroxypropyl-β-cyclodextrin IV (Experimental): Hydroxypropyl-β-cyclodextrin will be administered as Trappsol® Cyclo 25% (250mg/mL) by slow intravenous infusion over a period of 8 up to 9 hours.
  Interventions: Drug: Hydroxypropyl-β-cyclodextrin

INTERVENTIONS:
Drug: Hydroxypropyl-β-cyclodextrin — HP-β-CD will be administered as Trappsol® Cyclo 25% (250mg/mL) by slow intravenous infusion over a period of 8 up to 9 hours.
  Other Names: Hydroxypropyl-β-cyclodextrin (HP-β-CD); Trappsol® Cyclo

SUMMARY:
The purpose of this study is to provide continued access to treatment for NPC-1 after participation and completion of the Phase I trial CTD-TCNPC-101, when administered at doses of 1500 mg/kg and 2500 mg/kg by slow IV infusion over a period of 8 to 9 hours every two weeks.

DETAILED DESCRIPTION:
This is an open-label extension study of intravenous HP-β-CD (administered as Trappsol® Cyclo(TM)) in patients with NPC-1 to evaluate long-term safety and efficacy by providing continued access to treatment following completion of study CTD-TCNPC-101. Patients will receive medication at their home or local site under the supervision of a home nurse professional or at the parent site under the supervision of the site principal investigator. Patients will visit the parent site for safety and efficacy evaluations after receiving treatment for 3 months in the extension protocol.

Thereafter, visits to the parent site will be every 6 months until cessation. The study will continue until Trappsol® Cyclo (TM) becomes commercially available or study/site/patient discontinuation. All patients who complete study CTD-TCNCP-101 and pass the screening criteria will be eligible for this study. The study will be directed from parent site in the US. Vital signs, AEs Adverse Events (AEs) and concomitant meds will be recorded by the home nurse professional or deputy at the local site and reported immediately to the parent site for entry into the Electronic Data Capture (EDC) and reporting to the sponsor.

For logistical reasons home infusions will be permitted as long as AEs, infusion details and concomitants medications are reported directly to the parent site by an authorised deputy according to local guidelines. A Safety Review Committee (SRC) consisting of an independent advisor, the medical monitor, and the principal investigator will be established to review AEs and laboratory data throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Completion of study CTD-TCNPC-101 with no safety concerns at the final visit
* Negative urine pregnancy test for females of child bearing potential
* Patients must be legally resident in the USA with access to healthcare
* Written, informed consent

Exclusion Criteria:

* Inability to comply with the proposed protocol assessments or any uncertainty about their ability to give meaningful, informed consent (legal guardian may give consent with subject assent)
* Concurrent medical conditions representing a contraindication to any of the study medications
* Grade 3 renal impairment or worse as indicated by estimated Glomerular filtration rate (eGFR) < 60mL/min/1.73m2
* Clinical evidence of acute liver disease including symptoms of jaundice or right upper quadrant pain or International Normalised Ratio (INR) >1.8
* Male patients and female patients of childbearing potential who are not willing to use appropriate birth control (i.e. double barrier birth control) from enrollment until the follow-up visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2019-05-23 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs): Frequency, severity, time to onset, duration, and relatedness to study product | 1-104 weeks
  Adverse events (AEs): Frequency, severity, time to onset, duration, and relatedness to study product
Serious adverse events (SAEs): Frequency, severity, time to onset, duration and relatedness to study product | 1-104 weeks
  Serious adverse events (SAEs): Frequency, severity, time to onset, duration and relatedness to study product
Number of discontinuations due to AEs: Patient Discontinuation, Study Treatment Discontinuation, Study and Site Discontinuation | 1-104 weeks
  Discontinuation, Study and Site Discontinuation
Auditory capacity will be measured by behavioral auditory assessment | 1-104 weeks
  Auditory capacity will be measured by behavioral auditory assessment

SECONDARY OUTCOMES:
Change from baseline in total score as well as individual National Institute of Health (NIH) Niemann-Pick Disease Type C (NPC) Severity Scale (NCSS) | 1-104 weeks
  Change from baseline in total score as well as individual National Institute of Health (NIH) Niemann-Pick Disease Type C (NPC) Severity Scale (NCSS)

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Hastings, MD, Principal Investigator — UCSF Benioff Children's Hospital Oakland
Locations (1):
- UCSF Benioff Children's Hospital Oakland, Oakland, California, United States

REFERENCES:
- [Derived] Hastings C, Liu B, Hurst B, Cox GF, Hrynkow S. Intravenous 2-hydroxypropyl-beta-cyclodextrin (Trappsol(R) Cyclo) demonstrates biological activity and impacts cholesterol metabolism in the central nervous system and peripheral tissues in adult subjects with Niemann-Pick Disease Type C1: Results of a phase 1 trial. Mol Genet Metab. 2022 Dec;137(4):309-319. doi: 10.1016/j.ymgme.2022.10.004. Epub 2022 Oct 17. PMID 36279795